CLINICAL TRIAL: NCT05794490
Title: Continuous Learning to Increase Patient Safety - A Multi-method Study
Brief Title: Learning From Excellence in a Hospital Unit
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Gørill Birkeli, Principal Investigator, University Hospital, Akershus
Other Study IDs: 2022_3 and 2024_37
Record Dates: First submitted 2023-03-04; First posted 2023-04-03 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Health Personnel; Resilience; Patient Safety; Learning; Quality Improvement
Keywords: resilience; learning from excellence; healthcare quality improvement; safety culture; patient safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Learning from excellence — Health care professionals´ experiences of learning from excellence in a hospital unit

SUMMARY:
This study is based on the implementation of the method named "Learning-from-excellence", see methodology www.learningfromexcellence.com.

The project is a longitudinal cohort study based on data from both qualitative and quantitative data, presented in two different research articles, one qualitative and one quantitative, using :

* an electronic hosptal staff survey on "work-engagement, team collaboration, patient safety climate, and working conditions" before and after implementing Learning from Excellence.
* focus group interviews to explore experiences with the method of Learning from excellence from the view of healthcare professionals.

DETAILED DESCRIPTION:
One measure to improve patient safety, is to focus on improvements based on learning from errors (Safety-I). However, it is advocated that learning also should be based on situations where work goes well (Safety-II). Learning from Excellence (LfE) is an English initiative to learn from what works well and provide positive feedback to staff to increase resilience. LfE was implemented in a unit of a South-eastern Norwegian hospital trust between November 2022 and May 2023, using readily available resources from www.learningfromexcellence.com.

The qualitative data will be derived from five semi-structured focus group interviews, with nurses, physicians and change team representants. A descriptive design will be applied, and the data will be analysed using a more deductive, reflexive thematic analysis. Data from the focus group interviews will be taped on a recorder and stored at a secured computerised research place at Akershus University Hospital.

The gained knowledge from the focus group interviews in this study may provide in-depth knowledge on healthcare professionals' experiences in the novel field of learning from excellence, regarding the outcomes: learning, quality improvement work and resilience and culture in the workplace.

The quantitative part consist of aggregated data reports derived from the annual Norwegian hospital survey, which is a measure to explore connections between working environment, patient safety and Health-Environment-Safety in Norwegian hospitals, with a 5-point Likert response scale. From this report we derive answers from 20 questions, submittet before (March 2021 and 2022) and after (March 2023 and 2024), regarding the themes: Work engagement (n= 6), Team-collaboration (n=5) Patient safety climate (n=6) Working conditions (n=3). Thus, the study uses a longitudinal quasi-experimental pre-post intervention design, with a non-equivalent comparison unit.

The gained knowledge from the surveys may provide information if and how the method of Learning from excellence method impact the perceived:

* patient safety climate
* work engagement
* team-collaboration
* working conditions

ELIGIBILITY:
Inclusion Criteria Qualitative study:

* Nurses who had been working for at least six months on the premises
* Physicians who had either received or captured and reported peer excellence

Inclusion Criteria Quantitative study:

All nurses working on the premises who have answered questions in the annual hospital survey, between March 2021 and March 2024. Answers are collected on unit-level, not individual level.

Exclusion Criteria:

-

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The quantitative part of this longitudinal cohort study will collect data from all nurses working on the premises who have answered questions on the annual Norwegian hospital survey from March 2016 to March 2023.
  The qualitative part will include the aforementioned nurses, additionally, anaesthesiologists who have participated in the Learning from Excellence method.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Qualitative: Focus group interviews | 6 months after implementation of Learning from Excellence, i.e., May 2023
  Health care professionals´ experiences of learning from excellence in a hospital unit

SECONDARY OUTCOMES:
Quantitative: Survey from the nurses unit | From March 2021 to March 2024
  Aggregated data from the annual Norwegian hospital survey, which is a measure to explore connections between working environment, patient safety and Health-Environment-Safety in Norwegian hospitals

CONTACTS AND LOCATIONS:
Overall Officials: Anne Karin Lindahl, PhD, Study Director — University of Oslo Faculty of Medicine, Institute of Health and Society
Locations (1):
- Akershus University Hospital, Lørenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Birkeli G, Deilkas ECT, Ballangrud R, Lindahl AK. Implementing Learning from Excellence in a postanaesthesia care unit: a qualitative study of healthcare professionals' experiences after six months. BMC Health Serv Res. 2025 Apr 2;25(1):493. doi: 10.1186/s12913-025-12626-8. PMID 40176056